CLINICAL TRIAL: NCT00001057
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial of the Virologic Effect of Two Different Nucleoside Treatment Strategies (Zidovudine Versus Zidovudine in Combination With Didanosine) for HIV Infection in Subjects With CD4+ Counts >= 550 Cells/mm3
Brief Title: The Effectiveness of Two Anti-HIV Treatments in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 275; 11251 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To determine the effects of zidovudine (AZT) alone and in combination with didanosine (ddI) on viral load in the lymphoid tissue and blood of antiretroviral-naive, HIV-infected patients with CD4 counts greater than or equal to 550 cells/mm3.

Recent studies have shown that during the asymptomatic phase (clinical latency) of HIV infection, there is an extraordinarily large number of infected CD4+ lymphocytes and macrophages throughout the lymphoid system, both in latent and productive states. These findings support the belief that early intervention therapy with reverse transcriptase inhibitors could prolong the clinical latency period.

DETAILED DESCRIPTION:
Recent studies have shown that during the asymptomatic phase (clinical latency) of HIV infection, there is an extraordinarily large number of infected CD4+ lymphocytes and macrophages throughout the lymphoid system, both in latent and productive states. These findings support the belief that early intervention therapy with reverse transcriptase inhibitors could prolong the clinical latency period.

Patients are randomized to receive AZT alone, AZT plus ddI, or no therapy (placebo) daily for 48 weeks. Patients are followed at weeks 2, 4, and 8, and then every 8 weeks thereafter until week 48.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antibiotics for bacterial infections as clinically indicated.
* Recombinant erythropoietin (EPO) and G-CSF as clinically indicated for grade 3 or worse anemia and neutropenia, respectively.
* Antipyretics.
* Analgesics.
* Allergy medications.
* Oral contraceptives.
* Nonprescription medications such as vitamins or herbal therapies.

Concurrent Treatment:

Allowed:

* Radiation therapy to local lesion only.
* Acupuncture.

Patients must have:

* HIV seropositivity.
* CD4 count >= 550 cells/mm3.
* No ARC or AIDS conditions by CDC criteria.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Presence of factors predisposing to pancreatitis such as active alcoholism.
* Other medical conditions that would interfere with study compliance.

Concurrent Medication:

Excluded:

* Other antiretrovirals or systemic immunomodulators.
* Systemic corticosteroids.
* Systemic cytotoxic chemotherapy.
* Intravenous pentamidine.

Concurrent Treatment:

Excluded:

* Radiation therapy except to local lesion.

Patients with the following prior conditions are excluded:

* History of chronic diarrhea, defined as more than four loose or watery stools on average daily for the past month.
* History of grade 2 or worse peripheral neuropathy.
* History of pancreatitis.
* Bacterial infection requiring antibiotics within 14 days prior to study entry.

Prior Medication:

Excluded:

* Prior HIV therapy with antiretrovirals or systemic immunomodulators.

Prior Treatment:

Excluded within 2 weeks prior to study entry:

* Transfusion.

Active substance abuse or alcoholism.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105
Dates: Study Completion 1995-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erice A, Study Chair; Balfour H, Study Chair; Carey J, Study Chair; Henry K, Study Chair; Hasse A, Study Chair
Locations (7):
- United States (7):
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Case Western Reserve Univ, Cleveland, Ohio
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Univ of Texas Galveston, Galveston, Texas